CLINICAL TRIAL: NCT05506488
Title: Dasatinib and Quercetin, a Combination of Senolytics to Treat Fibrotic Non-alcoholic Fatty Liver Disease - the TRUTH Study
Brief Title: Dasatinib and Quercetin to Treat Fibrotic Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.0213
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: NAFLD; NASH With Fibrosis; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled proof-of-principle study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dasatinib plus Quercetin (Active Comparator): Day 0: (15 per arm, randomization). week 7: blood, fibroscan, ECG, questionnaires. week 14: blood, fibroscan, ECG, questionnaires. Week 21: blood, fibroscan, ECG, questionnaires, liver biopsy. end of study
  Interventions: Drug: Dasatinib 100 MG + Quercetin (1000 MG)
- placebo (Placebo Comparator): Day 0: (15 per arm, randomization). week 7: blood, fibroscan, ECG, questionnaires. week 14: blood, fibroscan, ECG, questionnaires. Week 21: blood, fibroscan, ECG, questionnaires, liver biopsy. end of study
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dasatinib 100 MG + Quercetin (1000 MG) — The intervention group will receive intermittent orally administered dasatinib (100 mg/day) plus quercetin (1000 mg/day) on three consecutive days for three consecutive weeks followed by a four-week medication free period. This cycle will be repeated three times.
  Arms: Dasatinib plus Quercetin
Other: Placebo — The placebo group will receive intermittent orally administered placebo tablets on three consecutive days for three consecutive weeks followed by a four-week medication free period. This cycle will be repeated three times.
  Arms: placebo

SUMMARY:
To examine the effect of dasatinib plus quercetin on liver fibrosis in individuals with biopsy proven NAFLD with fibrosis by performing a double-blind randomized controlled proof-of-principle study

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is estimated to affect approximately 25-30% of the population in Western countries and is now the leading cause of chronic liver disease globally. NAFLD is a progressive liver disease and approximately 30% of individuals progress from simple steatosis to Non-Alcoholic Steatohepatitis (NASH), which can further progress to cirrhosis and hepatocellular carcinoma. In the Netherlands, it is estimated that 2.5 million people have NAFLD and this number is thought to increase by 50% in the next 10 years driven by an increasing prevalence of obesity and type 2 diabetes, and an ageing population. Independent of other cardiometabolic diseases, cardiovascular disease is the leading cause of death in individuals with NAFLD, followed by extrahepatic malignancies and liver-related complications. NAFLD results in sustained healthcare costs and economic losses, and reduced health-related quality of life.

It is now widely accepted that liver fibrosis is a result of liver injury secondary to NAFLD and is a major predictor for liver-related and overall mortality in individuals with NAFLD. The process of fibrosis progression is not completely understood, and it can vary considerably from one individual to another. Several risk factors for fibrosis progression have been identified: age, hypertension, obesity and type 2 diabetes. As of to date, no treatment is available that proved to be successful to target hepatic fibrosis. The only therapeutic options currently available therefore are the control of the concomitant metabolic diseases in addition to diet and lifestyle changes. Unfortunately, this inevitably will lead to polypharmacy and thereby decreases treatment adherence and increases the risk of adverse events and interactions with other drugs.

Recently, cellular senescence has been put forward as a causal factor in the development and progression of NAFLD and NAFLD related liver fibrosis. Cellular senescence is one of the hallmarks of aging and is defined as a stable arrest of the cell cycle coupled to specific phenotypic changes. Senescent cells secrete a collection of proteins called the senescence-associated secretory phenotype (SASP). This pro-inflammatory secretome drives age-related tissue dysfunction. Interestingly, metabolic dysregulation is thought to favor cellular senescence in several tissues involved in the pathogenesis of NAFLD such as the liver, pancreas and adipose tissue, further perpetuating metabolic dysregulation. Of interest, cellular senescence can be targeted using senolytics. The combination of dasatinib, which is an EMA-approved tyrosine kinase inhibitor and the antioxidant quercetin, which is a flavonol present in many fruits and vegetables, successfully clears senescent cells. Recent work in humans and rodents have shown that tissue function, including liver metabolism, can be recovered by clearing senescent cells with senolytics including.

Due the potential role of senescence in NAFLD related fibrosis, dasatinib plus quercetin might thus be an interesting future therapeutic option to tackle NAFLD related fibrosis. Based on the long-term safety profile of these treatments and the high unmet clinical need as there currently is no treatment for NAFLD we aim to perform a double-blind randomized controlled proof-of-principle study in which patients with NAFLD related liver fibrosis will be treated with dasatinib plus quercetin intermittently three days per week for three weeks, followed by a four-week medication-free period. Subsequently, this treatment cycle will be repeated three times

ELIGIBILITY:
Inclusion Criteria:

Adult individuals, age > 18 years

* NAFLD with fibrosis score >2 according to the Steatosis Activity and Fibrosis score, but no cirrhosis histological diagnosis according to the SAF fibrosis score on a liver biopsy performed < 6 months before screening in the study and confirmed by central reading during the screening period.
* Individuals agrees to have a liver biopsy performed after the treatment
* Compensated liver disease with the following hematologic and biochemical criteria on entry into protocol:

  * ALAT <10x ULN
  * Hemoglobin > 11g/dL for females and 12 g/dL for males
  * White blood cell (WBC) > 2.5 K/ μL
  * Neutrophil count > 1.5 K μL
  * Platelets > 100 K/μL
  * Total bilirubin <35 μmol/L
  * Albumin >30 g/L
  * TP >80% or INR <1.4
  * Serum creatinine <1.3 mg/dL (men) or <1.1 mg/dL (women) or estimated glomerular filtration rate (eGFR) > 60mL/min/1.73m2
* Have a stable weight since the liver biopsy was performed defined by no more than a 5% loss of initial body weight
* Subjects should be able to give informed consent

Exclusion Criteria:

* Evidence of another form of liver disease
* History of sustained excess alcohol ingestion: daily consumption >30g/day (3 drinks per day) for males and >20 g/day (2 drinks per day) for females
* Unstable metabolic condition: weight change > 5 kg in the last three months, diabetes with poor glycaemic control (HbA1c > 8.5%), introduction of an antidiabetic or of an anti-obesity drug/malabsorptive or restrictive bariatric (weight loss) surgery in the past 6 months prior to screening
* Bariatric surgery
* ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose oestrogens, methotrexate, tetracycline or amiodarone in the previous 6 months
* Significant systemic or major illnesses other than liver disease, including congestive heart failure (class C and D of the AHA), unstable coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, organ transplantation, serious psychiatric disease, active malignancy, compromised immunity
* Pregnancy/lactation or inability to adhere to adequate contraception in woman of childbearing potential
* Body mass index (BMI) >45 kg/m2
* Type 1 diabetes
* Haemostasis disorders or current treatment with anticoagulants
* Contra-indication to liver biopsy
* History of/or current cardiac dysrhythmias and/or a history of cardiovascular disease event, including myocardial infarction, except patients with only well controlled hypertension
* QTc >450 msec on ECG
* Use of prescribed drugs dependent on CYP3A4 with narrow therapeutic window and strong inducers or inhibitors of CYP3A4
* Use of H2-antagonists and/or Proton Pump Inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the binary outcome improvement of fibrosis with at least 1-point without worsening of fibrosis and NAFLD score based on histology after 21 weeks (yes/no). Individuals will be labeled as responder or non-responder. | 21 week
  As assessed on the obtained liver biopsies before and after the treatment

SECONDARY OUTCOMES:
Mean change in number of senescent cells at baseline and end of treatment | 21 week
  As assessed on the obtained liver biopsies before and after the treatment
Percent of patients with reversal of NAFLD (Steatosis without ballooning and with or without mild inflammation) and no worsening of fibrosis) from baseline to end of treatment | 21 week
  As assessed on the obtained liver biopsies before and after the treatment
Global hepatic mRNA expression baseline to end of treatment | 21 week
  As assessed on the obtained liver biopsies before and after the treatment
Change in NAFLD activity score (NAS) | 21 week
  As assessed on the obtained liver biopsies before and after the treatment
change in Activity component of steatosis-activity-fibrosis (SAF) score: steatosis -1 point, lobular inflammation -1 point, ballooning -1 point | 21 week
  As assessed on the obtained liver biopsies before and after the treatment
change in Fibrosis-4 score (Fib-4 score) | 21 week
  Based on blood obtained before and after the treatment
Change in NAFLD Fibrosis Score (NFS) | 21 weeks
  Based on blood obtained before and after the treatment
Change in Liver enzymes | 21 weeks
  Based on blood obtained before and after the treatment
Change in Liver synthesis function | 21 weeks
  Based on blood obtained before and after the treatment
Change in liver stiffness and liver steatosis (with controlled attenuation parameter) measurement by Fibroscan | 21 weeks
  Based on Fibroscan scores obtained before and after the treatment
Change in Glycosylated haemoglobin type A1c (HbA1c) | 21 weeks
  Based on blood obtained before and after the treatment
Change in Fasting plasma glucose (FPG) | 21 weeks
  Based on blood obtained before and after the treatment
Change in Fasting glucagon | 21 weeks
  Based on blood obtained before and after the treatment
Change in Fasting insulin | 21 weeks
  Based on blood obtained before and after the treatment
change in Homeostatic model assessment of insulin resistance (HOMA-IR) | 21 weeks
  Based on blood obtained before and after the treatment
Change in RAND-36 questionnaires | 21 week
  Based on the questionnaires obtained before and after the treatment
Change in EQ-5D-5L questionnaires | 21 week
  Based on the questionnaires obtained before and after the treatment
Safety endpoints | 21 weeks
  * Number of treatment-emergent adverse events during the trial
  * Number of treatment-emergent myelosuppression
  * Number of treatment emergent infections
  * Number of subjects discontinuing treatment due to gastrointestinal adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No